CLINICAL TRIAL: NCT02565992
Title: Phase I Study of Intratumoral CAVATAK® (Coxsackievirus A21) and Pembrolizumab in Subjects With Advanced Melanoma (VLA-011 CAPRA)
Brief Title: Intratumoral CAVATAK (CVA21) and Pembrolizumab in Patients With Advanced Melanoma (VLA-011 CAPRA)
Acronym: CAPRA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Viralytics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V937-007; VLA-011 (Other: Viralytics Study ID)
Record Dates: First submitted 2015-09-30; First posted 2015-10-01 (Estimated); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Melanoma
Keywords: Pembrolizumab; Coxsackievirus A21; melanoma; CAVATAK; CVA21; checkpoint inhibitor
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab

ARMS (1):
- CAVATAK and pembrolizumab (Experimental): Intratumoral CAVATAK administration on trial days 1, 3, 5 and 8 and at 3-weekly intervals up to a maximum of 19 total with intravenous pembrolizumab (2 mg/kg solution) starting on day 8 and continuing every 3 weeks, up to 2 years.
  Interventions: Biological: CAVATAK; Drug: Pembrolizumab

INTERVENTIONS:
Biological: CAVATAK — Maximum dose of CVA21 is 3 x 10E+08 TCID50 (about 4.5 x 10E+06 TCID50/kg for a 70-kg patient) by intratumoral administration.
  Other Names: Coxsackievirus A21, CVA21
Drug: Pembrolizumab — Intravenous pembrolizumab at 2 mg/kg solution.

SUMMARY:
This study will employ a phase Ib design using the established dose of CAVATAK with pembrolizumab in subjects with advanced melanoma for whom pembrolizumab would be considered standard of care. Our hypothesis is that oncolysis of melanoma cells by CAVATAK will be important in amplifying the T-cell potentiating effects of pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with metastatic or unresectable stage IIIb/c of IV melanoma for whom treatment with pembrolizumab is indicated and who have at least one cutaneous, subcutaneous tumor or palpable lymph node amenable to intratumoral injection.
* At least one tumor must qualify to be an index lesion for modified WHO criteria.
* Subjects must have adequate hematologic, hepatic and renal function.
* ECOG performance status of 0 or 1.
* Anticipated lifespan greater than 12 weeks

Exclusion Criteria:

* Ocular primary tumors.
* Presence of any central nervous system tumor that has not been stable for at least 4 weeks off corticosteroids.
* Tumors lying in mucosal regions or close to an airway, major blood vessel or spinal cord.
* Subjects with active, known or suspected autoimmune or immunosuppressive disease.
* Subjects previously treated with CVA21.
* Subjects requiring systemic treatment with corticosteroids or other immunosuppressive medications within 14 days prior to the first treatment.
* Subject has received chemotherapy within the last 4 weeks prior to first treatment.
* Clinically significant cardiovascular disease.
* Females of childbearing potential must have negative serum or urine pregnancy test.
* Subjects requiring or using other investigational agents while on treatment in this trial.
* History of other malignancy within the last 3 years (with exceptions).
* Active infection requiring systemic therapy.
* Known history of HIV disease, active hepatitis B or hepatitis C.
* History or evidence of other clinically significant disorders that would pose a risk to subject safety.
* Inability to give informed consent and comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-12-17 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-04 (Actual)

PRIMARY OUTCOMES:
The incidence of dose-limiting toxicities (DLT) of intravenous pembrolizumab in combination with intratumoral CAVATAK will be assessed using CTCAE v. 4.0. | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - John Wayne Cancer Institute, Santa Monica, California
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Gabrail Cancer Center Research, Canton, Ohio

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Silk AW, O'Day SJ, Kaufman HL, Bryan J, Norrell JT, Imbergamo C, Portal D, Zambrano-Acosta E, Palmeri M, Fein S, Wu C, Guerreiro L, Medina D, Bommareddy PK, Zloza A, Fox BA, Ballesteros-Merino C, Ren Y, Shafren D, Grose M, Vieth JA, Mehnert JM. A phase 1b single-arm trial of intratumoral oncolytic virus V937 in combination with pembrolizumab in patients with advanced melanoma: results from the CAPRA study. Cancer Immunol Immunother. 2023 Jun;72(6):1405-1415. doi: 10.1007/s00262-022-03314-1. Epub 2022 Nov 29. PMID 36445410